CLINICAL TRIAL: NCT01842165
Title: The LuMEn Study: 177Lu-octreotate Treatment Outcome Prediction Using Multimodality Imaging in Refractory Neuroendocrine Tumours.
Brief Title: 177Lutetium-octreotate Treatment Prediction Using Multimodality Imaging in Refractory NETs
Acronym: LUMEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJBMNLUMEN; 2012-003666-41 (EudraCT Number)
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors
Keywords: Peptide Receptor Radionuclide Therapy (PRRT); Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 177Lu-octreotate therapy (Other): Treatment will consist of 177Lu-octreotate injections in fixed activities of 7,4 GBq (200 mCi) (±5%) each, given 12 weeks (±1 week) apart, injected intravenously simultaneously with nephroprotective perfusion of an amino acid solution.
  Interventions: Drug: Intravenous injection of 177Lu-octreotate

INTERVENTIONS:
Drug: Intravenous injection of 177Lu-octreotate — Treatment will consist of 177Lu-octreotate injections in fixed activities of 7,4 GBq (200 mCi) (±5%) each, given 12 weeks (±1 week) apart, injected intravenously simultaneously with nephroprotective perfusion of an amino acid solution.
  Other Names: 177Lu-DOTATATE; Lutate

SUMMARY:
The purpose of this study is to determine if 68Gallium-octreotate and 18Fluorodesoxyglucose uptake, apparent diffusion coefficient and post 177Lu-octreotate SPECT/CT dosimetry are reliable predictors for lesion-by-lesion treatment outcome.

DETAILED DESCRIPTION:
This is a feasibility study evaluating the use of 177Lutetium-octreotate in the treatment of advanced refractory Neuroendocrine Tumors.

Objectives of the study:

1. Primary (on a lesion basis): To assess the value of the following parameters (obtained through functional and molecular imaging) for predicting the lesion-by-lesion PRRT treatment outcome:

   * 18FDG uptake on 18FDG PET/CT
   * 68Ga-octreotate uptake on 68Ga-octreotate PET/CT
   * Apparent diffusion coefficient on diffusion weighted MRI (for these 3 parameters, absolute values at baseline)
   * Tumor dosimetry on post 177Lu-octreotate SPECT/CT after each cycle.
2. Secondary (on a patient basis): To generate a patient-based response model based on the previously defined parameters.
3. Exploratory (on a lesion basis): To assess the value of the parameters mentioned in the primary objective for predicting the lesion-by-lesion PRRT treatment outcome:

   * absolute values of the three imaging parameters and their relative changes after each cycle;
   * serial tumor dosimetry on post-177Lu-octreotate SPECT/CT after each cycle.

Treatment will consist of 177Lu-octreotate injections in fixed activities of 7,4 GigaBecqurel each, given 11-13 weeks apart, injected intravenously with simultaneous infusion of an amino acid solution. (Before amino acid nephroprotection, ondansetron, methylprednisolone and metoclopramid, are given intravenously in order to prevent nausea or vomiting). Approximately 30 min after the beginning of the amino acid solution, 177Lu-octreotate is co-infused over 15-30 minutes. The amino acid infusion is continued at the same rate for 3-5 more hours (total infusion lasts 4-6 hours).

In total, 4 cycles (= injections of 177Lu-octreotate) are planned. However, the total number of administered cycles will be limited by critical organ (kidneys and bone marrow) threshold toxicities.

Treatment efficacy will be assessed:

* on a lesion-basis (change of longest transversal diameter).
* on a patient-basis using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

ELIGIBILITY:
Inclusion Criteria:

Patient-based:

1. Age above or equal to 18 years.
2. Histology-proven advanced GEP-NETs.
3. Disease progression defined as follows (at least one of the following):

   - Radiological disease progression (according to RECIST 1.1) on an MRI or CT over the last 12 months Or

   - Disease progression on a somatostatin receptor-imaging, PET/CT or SPECT/CT over the last 12 months [apparition of new lesion(s) or increase in the transaxial plane diameter of more than 30% on the same imaging modality] Or

   - Both of the following criteria (a+b):
   1. clinical progression:

      * sustained (for more than 2 weeks) increase of NET-specific hormonal hypersecretion related symptom frequency by 50% or,
      * sustained (for more than 2 weeks) increase of severity by 1 grade (according to NCI-CTCAE version 4.03).
   2. biochemical progression: by increase of NET-specific tumor markers (plasma Chromogranin A, plasma NSE, urine 5-HIAA or other) in two successive measurements.
4. Disease refractory to SSA's and/or standard systemic therapy available in Belgium at the time of inclusion criteria.
5. Long-acting SSAs should be discontinued at least 4 weeks before study treatment start date and, if needed, switched to short-acting analogues which should be stopped 48h before the treatment date.
6. Adequate renal function with GFR ≥ 50 mL/min/1.73m2 (evaluated by 51Cr-EDTA test).
7. Adequate bone marrow function with hemoglobin ≥ 9 g/dL; neutrophil ≥ 1.5·103/μL; platelet count ≥ 100·103/μL.
8. Adequate liver function with total bilirubin ≤ 2 x ULN and transaminases ≤ 5 x ULN, serum albumin > 3 g/dL with normal prothrombin time (> 70%).
9. ECOG Performance Status ≤ 1.
10. Women of childbearing potential and men with partners of childbearing potential must agree to use a highly-effective form of contraception for the duration of study participation and up to six months after the end of the treatment. A pregnancy test (serum) must be performed within 4 weeks prior to inclusion for every female patient of childbearing potential and it must be negative.
11. Patient's written informed consent obtained prior to any study procedure.
12. All necessary baseline procedures should be performed within 4 weeks prior to first 177Lu-octreotate injection (D0).

    Lesion-based:
13. The patient must have at least one target lesion fulfilling all of the below criteria:

    * On the 68Ga-octreotate PET/CT: tumor uptake higher than the physiological liver uptake (grade III or IV of the Rotterdam visual score) in a lesion with longest transaxial plane diameter ≥20mm (measured on the CT, part of the PET/CT);
    * At least one of these lesions morphologically measurable according to RECIST 1.1 and progressive on the MRI (or CT if MRI is not applicable);
    * Target lesion should not have been previously irradiated.

Exclusion Criteria:

1. Resectable tumor with curative intent.
2. Any major surgery within the last 6 weeks prior to inclusion in the study
3. Radiotherapy, chemotherapy, embolization, mammalian target of rapamycin (mTOR)-inhibitors, receptor tyrosine-kinase inhibitors, interferon, or other investigational therapy within the last 12 weeks prior to inclusion in the study.
4. Diffuse bone marrow infiltration on the baseline 68Ga-octreotate PET/CT confirmed by MRI.
5. Prior external beam radiotherapy on kidneys or on more than 25% of bone marrow.
6. Patients with known uncontrolled brain metastases.
7. Patients with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the investigator's opinion, may interfere with completion of the study.
8. Pregnant or lactating patients.
9. Women of childbearing potential and men with partners of child-bearing potential refusing an adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05; Primary Completion 2022-01-14 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
The time to progression (TTP) for each target lesion assessed on MRI (or on CT scan if MRI is not possible). | 4 years [Anticipated]
  TTP is defined as the time between treatment initiation and objective tumor progression with censoring of patients who die as a result of any cause.

SECONDARY OUTCOMES:
Best morphological response according to RECIST 1.1 | 4 years [Anticipated]
Progression Free Survival | 4 years [Anticipated]
  PFS is defined as the time between treatment initiation and the first of the following events: disease progression (clinical or radiological) or death resulting from any cause.
Biochemical response (evolution of NET-specific tumoral uptake). | 4 years [Anticipated]

OTHER OUTCOMES:
The time to progression (TTP) for each target lesion assessed on MRI (or on CT scan if MRI is not applicable). | 4 years [Anticipated]

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flamen, M.D., Ph.D., Study Chair — Jules Bordet Institute; Amélie Deleporte, MD, Principal Investigator — Jules Bordet Institute; Alain Hendlisz, MD, Principal Investigator — Jules Bordet Institute; Ioannis Karfis, MD, Study Chair — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danieli R, Mileva M, Marin G, Kristanto P, Delbart W, Vanderlinden B, Wimana Z, Hendlisz A, Levillain H, Reynaert N, Flamen P, Karfis I. Evolution of dosimetric parameters through PRRT and potential impact on clinical practice: data from the prospective phase II LUMEN study. EJNMMI Res. 2024 Nov 18;14(1):110. doi: 10.1186/s13550-024-01163-w. PMID 39557730
- [Derived] Mileva M, Van Bogaert C, Marin G, Danieli R, Artigas C, Levillain H, Ameye L, Taraji-Schiltz L, Stathopoulos K, Wimana Z, Hendlisz A, Flamen P, Karfis I. 177 Lu-DOTATATE PRRT Safety and Organ-at-Risk Dosimetry in Patients With Gastroenteropancreatic Neuroendocrine Tumors : Data From the Prospective Phase 2 LUMEN Study. Clin Nucl Med. 2024 Sep 1;49(9):847-853. doi: 10.1097/RLU.0000000000005330. Epub 2024 Jun 19. PMID 38914016
- [Derived] Mileva M, Marin G, Levillain H, Artigas C, Van Bogaert C, Marin C, Danieli R, Deleporte A, Picchia S, Stathopoulos K, Jungels C, Vanderlinden B, Paesmans M, Ameye L, Critchi G, Taraji-Schiltz L, Velghe C, Wimana Z, Bali M, Hendlisz A, Flamen P, Karfis I. Prediction of 177Lu-DOTATATE PRRT Outcome Using Multimodality Imaging in Patients with Gastroenteropancreatic Neuroendocrine Tumors: Results from a Prospective Phase II LUMEN Study. J Nucl Med. 2024 Feb 1;65(2):236-244. doi: 10.2967/jnumed.123.265987. PMID 38164576